CLINICAL TRIAL: NCT07135388
Title: Treatment of Sarcopenia With Food for Special Medical Purposes in Rheumatologic Patients
Brief Title: Treatment of Rheumatologic Patients With Sarcopenia
Acronym: REU-SA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Michele Barone, Associate Professor, University of Bari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol # 0084855/06/11/2020; Study # 6557 (Other: Policlinic University Hospital local ethics committee)
Record Dates: First submitted 2025-08-03; First posted 2025-08-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Rheumatic Diseases
Keywords: Sarcopenia; Rheumatologic diseases; Food for Special Medical Purposes
MeSH Terms: conditions — Rheumatic Diseases; Sarcopenia | interventions — Food

STUDY DESIGN:
Intervention Model Description: Patients were evaluated before starting the nutritional treatment, and three months later.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rheumatologic sarcopenic patients receiving high protein, high content of HMB oral supplement (Other): Patients received for three months an oral supplementation with a protein supplement high in branched-chain amino acids and β-hydroxy-β-methyl-butyrate (HMB)
  Interventions: Dietary Supplement: Food for special medical purposes

INTERVENTIONS:
Dietary Supplement: Food for special medical purposes — Oral supplementation with a protein supplement high in branched-chain amino acids and β-hydroxy-β-methyl-butyrate (HMB)

SUMMARY:
Sarcopenia is defined as a pathological condition related to muscle strength and muscle mass reduction. It is caused by ageing (primary sarcopenia) and diseases associated with systemic inflammation (secondary sarcopenia). Systemic inflammation in rheumatological diseases often leads to physical inactivity, which is the main predictor of sarcopenia in this pathological condition. In these patients, the treatment of sarcopenia must necessarily include an appropriate nutritional approach, and the addition of oral supplements should be considered a complementary approach.

DETAILED DESCRIPTION:
Sarcopenia is linked to two distinct pathogenetic mechanisms that often overlap: ageing (primary sarcopenia), and diseases associated with either systemic inflammation or impaired physical activity, or nutritional deficiencies (secondary sarcopenia). Some of the latter mechanisms are intimately connected since the pathway to sarcopenia often begins with a chronic disease that triggers systemic inflammation, leading to physical inactivity, as occurs in rheumatological diseases. Notably, in these patients, the reduction in physical activity leading to sarcopenia represents a prognostic indicator for potential complications and compromised quality of life.

Skeletal muscle trophism is influenced by hormone-like factors known as myokines, which are mainly secreted by muscles themselves, and by cytokines. Among these molecules, irisin, decorin, myonectin, myostatin, and interleukin-15 have been widely studied to develop pharmacological strategies to counteract sarcopenia.

In any case, the treatment of sarcopenia must necessarily include an appropriate nutritional approach that should consider both specific dietary components (dietary patterns) and nutrient intakes (total calories). As a matter of fact, specific dietary patterns are increasingly considered in nutritional studies on sarcopenia.

Currently, it has been observed that "high-quality diets" are associated with better physical functionality and a reduced risk of sarcopenia. However, although some nutrients and dietary patterns seem to have a potential protective effect against sarcopenia, in the presence of pathological conditions, the addition of oral nutritional supplements should offer the opportunity of adding high levels of specific nutritional components which are able to promote muscle trophism.

In this prospective longitudinal study, we evaluated the effect of a specific food for special medical purposes (FSMPs) supplementation on muscle strength, muscle mass, and muscle quality in rheumatologic patients with sarcopenia. In addition, we assessed myokine and cytokine variations in the serum, which are associated with this nutritional approach.

ELIGIBILITY:
Inclusion Criteria: Rheumatologic patients able to perform the handgrip test.

Exclusion Criteria: Upper limb arthropathy, chronic kidney disease with an eGFR <50 ml/min, severe congestive heart failure, cancer, decompensated diabetes, severe respiratory failure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle mass | The interval between the beginning and the end of the single treatment was three months.
  Muscle mass was assessed at time zero and after three months of oral supplementation by bioimpedance analysis
Muscle strength | The interval between the beginning and the end of the single treatment was three months
  Muscle strength was assessed at time zero and after three months of oral supplementation by a dynamometer

SECONDARY OUTCOMES:
Assessment of myokines and cytokines blood levels | The interval between the blood collection performed at the beginning and the end of the single treatment was three months
  Blood was collected at time zero and after three months of oral supplementation to evaluate some myokines (irisin, DBNF, decorin, myostatin) and IL-15.

CONTACTS AND LOCATIONS:
Overall Officials: Michele BARONE, Associate Professor, Principal Investigator — University of Bari
Locations (1):
- Polyclinic University Hospital, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: Undecided
I will share data upon formal request by other researchers.

REFERENCES:
- [Background] Barone M, Viggiani MT, Anelli MG, Fanizzi R, Lorusso O, Lopalco G, Cantarini L, Di Leo A, Lapadula G, Iannone F. Sarcopenia in Patients with Rheumatic Diseases: Prevalence and Associated Risk Factors. J Clin Med. 2018 Dec 1;7(12):504. doi: 10.3390/jcm7120504. PMID 30513782